CLINICAL TRIAL: NCT04063826
Title: Pilot Study to Assess PET-MR Imaging for the Detection and Quantitation of Early Fibrosis in Patients With Steatohepatitis and Chemotherapy-associated Steatohepatitis in Hepatic Metastatic Disease
Brief Title: PET-MR Study of Fatty Liver
Acronym: iDOSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17HH3944
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Steatohepatitis
Keywords: PET MR Imaging; Steatohepatitis; Chemotherapy associated steatohepatitis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Intervention Model Description: In the first part 3 patients will be imaged, 2 with severe biopsy proven SH and one with severe CASH. Thereafter, depending on the imaging results, the second part will include up to 7 patients with mild to moderate SH and those with mild to moderate CASH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET MRI Scan (Other): Imaging scan of the liver
  Interventions: Device: PET MRI

INTERVENTIONS:
Device: PET MRI — All participants will have a liver scan

SUMMARY:
This is a pilot, translational study designed to explore the feasibility of molecular imaging with FBA-A20FMDV2, radiolabelled with fluorine-18 ([18F]-FBA-A20FMDV2), in patients with SH and CASH in hepatic metastatic disease. FBA-A20FMDV2, a synthetic peptide derived from the foot and mouth disease virus (FMDV), has been shown pre-clinically to specifically bind to the epithelial specific integrin αvβ6 which is known to be overexpressed in tumours. In this study, we aim to evaluate the uptake of [18F]-FBA-A20FMDV2 ([18F]-IMAFIB) in patients with SH and CASH in CRC hepatic metastatic disease using PET. Up to ten subjects will undergo [18F]-FBA-A20FMDV-PET scanning. An adaptive study design will enable us to determine the optimal imaging protocol for future studies.

DETAILED DESCRIPTION:
This is a pilot study in two parts that aims to determine the feasibility of conducting PET-MR imaging using [18F]-FBA-A20FMDV2 ([18F]-IMAFIB) and novel PET-MR imaging in patients with SH and CASH in CRC hepatic metastatic disease. A combination of factors will be used to determine the feasibility of [18F]-IMAFIB PET-MR imaging including visual adequacy of the PET-MR image, adequate signal to noise ratio and the ability to evaluate changes in [18F]-IMAFIB uptake and PET-MR parameters. In addition, the operational feasibility of this study will be assessed. Up to 10 patients will be evaluated in this study. The number of patients to be included in this heterogeneous cohort of patients has been based on feasibility considerations taking into account recruitment rates and not on any formal statistical evaluation. An adaptive study design will be used with patients with imaging results being continuously assessed. In the first part 3 patients will be imaged, 2 with severe biopsy proven SH and one with severe CASH. Thereafter, depending on the imaging results, the second part will include up to 7 patients with mild to moderate SH and those with mild to moderate CASH. If there are major changes in the imaging protocol an amendment to the ethics committee will be submitted.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent prior to admission to this study.
* Female or male aged ≥18 years.
* Patients with clinical or histological diagnosis of SH or CASH, having received neoadjuvant chemotherapy for CRC hepatic metastatic disease prior to hepatic resection.
* Female patients of childbearing potential or male patients with female partners of child-bearing potential must agree to use adequate contraception as described in the protocol from the day of the scan and until 4 weeks after the scan.
* Negative urine pregnancy test for female patients of childbearing potential performed on the day of the PET Scan.

Exclusion Criteria:

* Breast feeding or pregnant women female patients.
* Previous or current exposure to animals that may harbour the FMDV.
* Previous long-term (≥ 3 months) residence in a country where FMDV is endemic (most parts of Africa, Middle East, Asia and parts of South America; see Appendix 1).
* Participant feels unable to lie flat on their back for a period of up to 95 minutes in the scanner.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of the tracer, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
* Contraindications to MRI scanning (as assessed by MRI safety questionnaire) which include, but are not limited to:

  1. Intracranial aneurysm clips or other metallic objects.
  2. History of intra-orbital metal fragments that have not been removed by a medical professional.
  3. Pacemakers, or other implanted cardiac rhythm management devices and non-MR compatible heart valves.
  4. Inner ear implants.
* Patients who have been involved in another research study within the last 30 days.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of [18F]-IMAFIB expressed as standardised uptake value (SUV) | 9 months
  To evaluate the feasibility of [18F]-IMAFIB-PET imaging in patients with hepatic metastatic disease

SECONDARY OUTCOMES:
Time Activity Curves (TACs) of [18F]-IMAFIB and the | 9 months
  The find the optimal PET scan time

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Spalding, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No